CLINICAL TRIAL: NCT01635244
Title: Trifecta Comparative Stress Hemodynamic Study (Randomized Comparison of Exercise Hemodynamics and Left Ventricular Remodeling With Aortic Bioprostheses After Aortic Valve Replacement for Aortic Stenosis)
Brief Title: Hemodynamic Comparison of Tissue Aortic Valves
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, David Bach, MD, Professor of Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N015029-00
Record Dates: First submitted 2012-07-01; First posted 2012-07-09 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2016-12

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic valve prosthesis; Aortic valve hemodynamics; Prosthesis-patient mismatch; Left ventricular diastolic function; Left ventricular remodeling
MeSH Terms: conditions — Aortic Valve Stenosis; Ventricular Remodeling | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Freestyle (Active Comparator): Aortic valve replacement will be performed with a Freestyle stentless aortic bioprosthesis (Medtronic Cardiovascular; Minneapolis, MN).
  Interventions: Device: Aortic valve replacement
- Magna Ease (Active Comparator): Aortic valve replacement will be performed with a Magna Ease aortic bioprosthesis (Edwards Lifesciences; Irvine, CA).
  Interventions: Device: Aortic valve replacement
- Trifecta (Active Comparator): Aortic valve replacement will be performed with a Trifecta aortic bioprosthesis (St. Jude Medical; St. Paul, MN).
  Interventions: Device: Aortic valve replacement

INTERVENTIONS:
Device: Aortic valve replacement — Clinically indicated aortic valve replacement will be performed using one of three approved tissue valves (Freestyle, Magna Ease, or Trifecta).

SUMMARY:
The purpose of this study is to:

1. Assess for hemodynamic differences at rest and with exercise between three clinically available tissue aortic valves.
2. Assess for differences in left ventricular (LV) reverse remodeling (recovery of LV hypertrophy, and changes in LV systolic and diastolic function) after aortic valve replacement for severe aortic stenosis (AS) between three clinically available aortic valve bioprosthesis.

DETAILED DESCRIPTION:
Various aortic valve prostheses have unique hemodynamic characteristics, and there is on-going interest in defining those hemodynamic characteristics in the interest of avoiding residual LV outflow obstruction and prosthesis-patient mismatch (residual LV outflow obstruction despite a normally functioning prosthesis ) after aortic valve replacement. Attempts to compare hemodynamics between prostheses have been limited by different sizing systems used by various manufacturers (precluding meaningful comparison of valves by valve size) and biological variability of in vivo gradients and effective orifice area for any valve (making potentially small differences in hemodynamics difficult to detect). Assessment of hemodynamics during increased cardiac output associated with exercise testing has been used to better define potentially subtle differences in hemodynamics between valve prostheses. In addition, assessment for change in LV geometry (notably including LV hypertrophy) after aortic valve replacement has been used as a surrogate marker of aortic prosthesis hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Severe aortic stenosis (AS) based on overall clinical impression, with or without aortic valve mean gradient ≥ 40 mm Hg, EOA < 1.0 cm2, or EOA index < 0.6 cm2/m2.
* Scheduled for clinically indicated elective aortic valve replacement for a primary diagnosis of severe AS.
* Less than moderate aortic regurgitation on preoperative testing.
* Isolated aortic valve replacement; or aortic valve replacement with concomitant coronary artery bypass grafting, ascending aorta repair, or mitral and/or tricuspid annuloplasty for functional mitral regurgitation / tricuspid regurgitation.
* Left ventricular ejection fraction ≥ 40% on preoperative testing.
* Physically able and willing to pedal a recumbent bicycle.
* Patient and surgeon agree that the patient will undergo valve replacement with a bioprosthesis.
* Patient and surgeon agree that the use of one specific bioprosthesis manufacturer / model is not indicated based on clinical criteria.
* Willing to undergo randomization to have implanted one of three bioprosthesis at the time of aortic valve replacement.
* Willing and able to undergo preoperative echocardiography/Doppler for purposes of the research study.
* Willing and able to undergo post-operative exercise stress echocardiography/Doppler 5 to 7 months after valve replacement for purposes of the research protocol.

Exclusion Criteria:

* Age < 18 years.
* AS felt by overall clinical impression to be less than severe.
* Aortic valve replacement is urgent or emergent.
* Moderate of more aortic regurgitation on preoperative testing.
* Concomitant mitral or tricuspid valve replacement.
* Left ventricular ejection fraction < 40% on preoperative testing.
* Physically unable or unwilling to pedal a recumbent bicycle.
* Planned aortic valve replacement with a mechanical prosthesis.
* Operating surgeon believes that any one of the three protocol bioprosthetic devices is contraindicated based on clinical criteria.
* Not willing to undergo randomization to have implanted one of three bioprosthesis.
* Unwilling or unable to undergo preoperative echocardiography/Doppler for purposes of the research protocol.
* Unwilling or unable to undergo post-operative exercise stress echocardiography/Doppler 5 to 7 months after valve replacement for purposes of the research protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Bach, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health Systems, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Bach DS, Patel HJ, Kolias TJ, Deeb GM. Randomized comparison of exercise haemodynamics of Freestyle, Magna Ease and Trifecta bioprostheses after aortic valve replacement for severe aortic stenosis. Eur J Cardiothorac Surg. 2016 Aug;50(2):361-7. doi: 10.1093/ejcts/ezv493. Epub 2016 Jan 27. PMID 26819292

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Freestyle | Magna Ease | Trifecta
Started | 18 | 22 | 20
Completed | 17 | 21 | 18
Not Completed | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Freestyle | Magna Ease | Trifecta | Total
Number analyzed (Participants) | 17 | 21 | 18 | 56
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 74 [64 to 80] | 67 [61 to 74] | 71 [64 to 76] | 70 [63 to 78]
Gender [Count of Participants; unit: Participants]
  Female | 6 | 9 | 4 | 19
  Male | 11 | 12 | 14 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 21 | 17 | 54
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 16 | 21 | 17 | 54
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 17 | 21 | 18 | 56

OUTCOME MEASURES:

1. Primary Outcome: Aortic Valve Mean Gradient (mm Hg) at Peak Exercise
Description: This is a measure of the resistance to flow across the aortic bioprosthesis.
Time Frame: 6 months after aortic valve replacement
Measure: Median (Inter-Quartile Range); unit: mm Hg
Arm/Group | Freestyle | Magna Ease | Trifecta
Number analyzed (Participants) | 17 | 21 | 18
mm Hg | 11 [8 to 16] | 14 [11 to 17] | 11 [8 to 13]

ADVERSE EVENTS:
Arm/Group | Freestyle | Magna Ease | Trifecta
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/18 | 0/22 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No